CLINICAL TRIAL: NCT03632083
Title: A Range of Contact Lenses and Care System Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C17-635 (EX-MKTG-95)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Contact Lens Solutions

STUDY DESIGN:
Intervention Model Description: This is a double-masked, randomized, contralateral, crossover study design. Lenses are worn as an unmatched pair.
Who Masked: Participant, Investigator
Masking Description: The first solution, the randomisation determines that the right lens will wear the fanfilcon A lens and the left eye will wear the comfilcon A lens for two hours of wear, with a two-day 'wash-out' period and the laterality of the lenses will be swapped for the second solution for two hours of wear. Lenses will be provided in lens cases which do not detail lens or care system information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hy-Care Contact Lens Solution (Active Comparator): Each subject will wear fanfilcon A soft contact lens in one eye and comfilcon A soft contact lens in the other eye with each lens having been soaked overnight in the Hy-Care contact lens solution.
  Interventions: Device: Hy-Care Contact Lens Solution; Device: fanfilcon A soft contact lens; Device: comfilcon A soft contact lens
- Lite Contact Lens Solution (Active Comparator): Each subject will wear fanfilcon A soft contact lens in one eye and comfilcon A soft contact lens in the other eye with each lens having been soaked overnight in the Lite contact lens solution.
  Interventions: Device: Lite Contact Lens Solution; Device: fanfilcon A soft contact lens; Device: comfilcon A soft contact lens

INTERVENTIONS:
Device: Hy-Care Contact Lens Solution — Hy-Care Contact Lens Solution
  Arms: Hy-Care Contact Lens Solution
Device: Lite Contact Lens Solution — Lite Contact Lens Solution
  Arms: Lite Contact Lens Solution
Device: fanfilcon A soft contact lens — fanfilcon A soft contact lens
Device: comfilcon A soft contact lens — comfilcon A soft contact lens

SUMMARY:
The objective of this study is to compare the short-term clinical response to all combinations of two lens types: fanfilcon A and comfilcon A with two care systems: Hy-Care and Lite. The primary variables of interest are short-term biomicroscopy signs. Other variables of interest include subjective response and visual performance.

DETAILED DESCRIPTION:
Subjects were randomized to wear fanfilcon A soft contact lens in one eye and comfilcon A soft contact lens in the other eye with each lens having been soaked overnight in the Hy-Care contact lens solution and Lite contact lens solution.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (18) and capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They agree not to participate in other clinical research for the duration of this study.
5. They can be satisfactorily fitted with the study lens for a period of approximately 2 hours.
6. They can attain at least 0.20 logMAR distance high contrast visual acuity in each eye with their habitual spectacles.
7. They currently wear daily disposable soft contact lenses or have done so in the previous six months.
8. They are willing to comply with the wear schedule (approximately 2 hours on two different days)
9. They own a wearable pair of spectacles and agree to bring these to study visits.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They currently wear reusable soft contact lenses in both eyes.
4. They are using any topical medication such as eye drops or ointment.
5. They have had cataract surgery.
6. They have had corneal refractive surgery.
7. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
8. They are pregnant or breast-feeding.
9. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
10. They have Type 2 or greater corneal staining prior to lens application at Visit 1 or 2
11. They have corneal staining covering greater than 20% in any corneal region at Visit 1a or 2a
12. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
13. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD MCOptom FAAO FBCLA, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-masked, contralateral, cross-over study in which subjects were randomized to wear fanfilcon A soft contact lens in one eye and comfilcon A soft contact lens in the other eye with each lens having been soaked overnight in a lens care product Lite or Hy-Care.
Units Other Than Participants: Eyes
Groups:
- Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Right Eye: Subjects were randomized to wear comfilcon A lens soaked overnight in the Hy-Care solution on the right eye for two hours then wear fanfilcon A lens soaked overnight in the Lite Solution on right eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Hy-Care - Fanfilcon A Then Lite - Comilcon A on Left Eye: Subjects were randomized to wear fanfilcon A lens soaked overnight in the Hy-Care solution on the left eye for two hours then wear comfilcon A lens soaked overnight in the Lite Solution on left eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Hy-Care - Fanfilcon A Then Lite - Comfilcon A on Right Eye: Subjects were randomized to wear fanfilcon A lens soaked overnight in the Hy-Care solution on the right eye for two hours then wear comfilcon A lens soaked overnight in the Lite Solution on right eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Left Eye: Subjects were randomized to wear comfilcon A lens soaked overnight in the Hy-Care solution on the left eye for two hours then wear fanfilcon A lens soaked overnight in the Lite Solution on left eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Right Eye: Subjects were randomized to wear comfilcon A lens soaked overnight in the Lite solution on the right eye for two hours then wear fanfilcon A lens soaked overnight in the Hy-Care Solution on right eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Left Eye: Subjects were randomized to wear fanfilcon A lens soaked overnight in the Lite solution on the left eye for two hours then wear comfilcon A lens soaked overnight in the Hy-Care Solution on left eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Right Eye: Subjects were randomized to wear fanfilcon A lens soaked overnight in the Lite solution on the right eye for two hours then wear comfilcon A lens soaked overnight in the Hy-Care solution on right eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
- Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Left Eye: Subjects were randomized to wear comfilcon A lens soaked overnight in the Lite solution on the left eye for two hours then wear fanfilcon A lens soaked overnight in the Hy-Care Solution on left eye for 2 hours.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Lite Contact Lens Solution: Lite Contact Lens Solution comfilcon A soft contact lens: comfilcon A soft contact lens fanfilcon A soft contact lens: fanfilcon A soft contact lens
Period: First Intervention
Arm/Group | Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Right Eye | Hy-Care - Fanfilcon A Then Lite - Comilcon A on Left Eye | Hy-Care - Fanfilcon A Then Lite - Comfilcon A on Right Eye | Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Left Eye | Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Right Eye | Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Left Eye | Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Right Eye | Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Left Eye
Started | 5; 5 Eyes | 5; 5 Eyes | 7; 7 Eyes | 7; 7 Eyes | 9; 9 Eyes | 9; 9 Eyes | 7; 7 Eyes | 7; 7 Eyes
Completed | 5; 5 Eyes | 5; 5 Eyes | 7; 7 Eyes | 7; 7 Eyes | 9; 9 Eyes | 9; 9 Eyes | 7; 7 Eyes | 7; 7 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes
Period: Second Intervention
Arm/Group | Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Right Eye | Hy-Care - Fanfilcon A Then Lite - Comilcon A on Left Eye | Hy-Care - Fanfilcon A Then Lite - Comfilcon A on Right Eye | Hy-Care - Comfilcon A Then Lite - Fanfilcon A on Left Eye | Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Right Eye | Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Left Eye | Lite - Fanfilcon A Then Hy-Care - Comfilcon A on Right Eye | Lite - Comfilcon A Then Hy-Care - Fanfilcon A on Left Eye
Started | 5; 5 Eyes | 5; 5 Eyes | 7; 7 Eyes | 7; 7 Eyes | 9; 9 Eyes | 9; 9 Eyes | 7; 7 Eyes | 7; 7 Eyes
Completed | 5; 5 Eyes | 5; 5 Eyes | 7; 7 Eyes | 7; 7 Eyes | 9; 9 Eyes | 9; 9 Eyes | 7; 7 Eyes | 5; 5 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes | 2; 2 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Subjects were randomized to wear fanfilcon A soft contact lens in one eye and comfilcon A soft contact lens in the other eye with each lens having been soaked overnight in the Hy-Care contact lens solution and Lite contact lens solution.
  Contact Lens Solution: Hy-Care Contact Lens Solution Contact Lens Solution: Lite contact lens solution
Arm/Group | Overall Participants
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Biomicroscopy - Conjuctival Hyperaemia
Description: Ocular physiology assessment of fanfilcon A and comfilcon A contact lenses with lens care products Lite and Hy-Care biomicroscopy (Scale 0-4, 0.25 steps, 0=normal, 4=severe).
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Hy-Care Contact Lens Solution - Comfilcon A: Each subject will wear comfilcon A soft contact lens in one eye with lens having been soaked overnight in the Hy-Care contact lens solution.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Contact lens: comfilcon A soft contact lens
- Hy-Care Contact Lens Solution - Fanfilcon A: Each subject will wear fanfilcon A soft contact lens in one eye with lens having been soaked overnight in the Hy-Care contact lens solution.
  Contact Lens Solution: Hy-Care Contact Lens Solution
  contact lens: fanfilcon A soft contact lens
- Lite Contact Lens Solution - Comfilcon A: Each subject will wear comfilcon A soft contact lens in one eye with lens having been soaked overnight in the Lite contact lens solution.
  Contact Lens Solution: Lite Contact Lens Solution
  Contact lens: comfilcon A soft contact lens
- Lite Contact Lens Solution - Fanfilcon A: Each subject will wear fanfilcon A soft contact lens in one eye with lens having been soaked overnight in the Lite contact lens solution.
  Contact Lens Solution: Lite contact Lens Solution
  Contact lens: fanfilcon A soft contact lens
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.95 (0.22) | 0.94 (0.23) | 0.91 (0.23) | 0.91 (0.21)

2. Primary Outcome: Biomicroscopy - Conjuctival Hyperaemia
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 1.01 (0.21) | 1.01 (0.21) | 0.99 (0.24) | 0.99 (0.25)

3. Primary Outcome: Biomicroscopy - Limbal Hyperaemia
Description: as for outcome 1
Time Frame: Baseline (before contact lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.86 (0.26) | 0.85 (0.28) | 0.76 (0.30) | 0.76 (0.28)

4. Primary Outcome: Biomicroscopy - Limbal Hyperaemia
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.90 (0.27) | 0.90 (0.28) | 0.81 (0.29) | 0.81 (0.31)

5. Primary Outcome: Biomicroscopy - Corneal Vascularisation
Description: as for outcome 1
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Groups:
- Hy-Care Contact Lens Solution - Comfilcon A: Each subject will wear comfilcon A soft contact lens in one eye with each lens having been soaked overnight in the Hy-Care contact lens solution.
  Hy-Care Contact Lens Solution: Hy-Care Contact Lens Solution Contact lens: comfilcon A soft contact lens
- Lite Contact Lens Solution - Comfilcon A: Each subject will wear comfilcon A soft contact lens in one eye with each lens having been soaked overnight in the Lite contact lens solution.
  Contact Lens Solution: Lite Contact Lens Solution
  Contact lens: comfilcon A soft contact lens
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.08 (0.15) | 0.08 (0.15) | 0.06 (0.12) | 0.06 (0.12)

6. Primary Outcome: Biomicroscopy - Corneal Vascularisation
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.09 (0.17) | 0.09 (0.17) | 0.06 (0.12) | 0.05 (0.12)

7. Primary Outcome: Biomicroscopy - Microcysts
Description: as for outcome 1
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

8. Primary Outcome: Biomicroscopy - Microcysts
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

9. Primary Outcome: Biomicroscopy - Oedema
Description: as for outcome 1
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

10. Primary Outcome: Biomicroscopy - Oedema
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

11. Primary Outcome: Biomicroscopy - Conjunctival Staining
Description: as for outcome 1
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 0.30 (0.32) | 0.34 (0.32) | 0.33 (0.30) | 0.33 (0.32)

12. Primary Outcome: Biomicroscopy - Conjunctival Staining
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 1.00 (0.50) | 0.91 (0.43) | 1.16 (0.41) | 1.09 (0.44)

13. Primary Outcome: Biomicroscopy - Papillary Conjunctivitis
Description: as for outcome 1
Time Frame: Baseline (before lens insertion)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 1.08 (0.27) | 1.06 (0.27) | 1.09 (0.27) | 1.08 (0.28)

14. Primary Outcome: Biomicroscopy - Papillary Conjunctivitis
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 1.10 (0.27) | 1.08 (0.27) | 1.08 (0.28) | 1.07 (0.25)

15. Secondary Outcome: Comfort
Description: Subjective ratings of comfort for each pair of lenses (scale: 0-100; 0=Cannot be tolerated,100=Cannot be felt).
Time Frame: Baseline 5 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 88.2 (11.8) | 93.5 (7.2) | 90.0 (12.4) | 90.8 (9.0)

16. Secondary Outcome: Comfort
Description: Subjective ratings of comfort for each pair of lenses (scale: 0-100; 0=Cannot be tolerated,100=Cannot be felt).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 90.5 (10.2) | 89.9 (13.0) | 92.3 (10.8) | 92.0 (11.6)

17. Secondary Outcome: Dryness
Description: Subjective ratings of dryness for each pair of lenses measured only at follow up (scale: 0-100; 0=Intolerable levels of dryness, 100=No sensation of dryness).
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 92.6 (7.7) | 90.3 (12.5) | 91.5 (12.5) | 91.7 (12.0)

18. Secondary Outcome: Overall Score
Description: Subjective ratings of overall score for each pair of lenses (scale: 0-100; 0=Cannot use lenses, 100=Highly impressed with lenses overall).
Time Frame: Baseline 5 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 89.0 (13.4) | 90.8 (12.2) | 92.2 (8.2) | 92.0 (8.3)

19. Secondary Outcome: Overall Score
Description: as for outcome 18
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
Number analyzed (Participants) | 28 | 28 | 28 | 28
Number analyzed (Eyes) | 28 | 28 | 28 | 28
units on a scale | 90.3 (9.4) | 89.1 (11.8) | 91.4 (12.4) | 87.1 (19.7)

ADVERSE EVENTS:
Time Frame: From baseline to follow up visit for an average of 2 hours, up to maximum of 14 days.
Groups:
- Hy-Care Contact Lens Solution - Comfilcon A: Contact Lens Solution: Hy-Care Contact Lens Solution Contact lens: comfilcon A soft contact lens
- Hy-Care Contact Lens Solution - Fanfilcon A: Contact Lens Solution: Hy-Care Contact Lens Solution
  contact lens: fanfilcon A soft contact lens
- Lite Contact Lens Solution - Comfilcon A: Contact Lens Solution: Lite Contact Lens Solution
  Contact lens: comfilcon A soft contact lens
- Lite Contact Lens Solution - Fanfilcon A: Contact Lens Solution: Lite contact Lens Solution
  Contact lens: fanfilcon A soft contact lens
Arm/Group | Hy-Care Contact Lens Solution - Comfilcon A | Hy-Care Contact Lens Solution - Fanfilcon A | Lite Contact Lens Solution - Comfilcon A | Lite Contact Lens Solution - Fanfilcon A
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT03632083/Prot_SAP_000.pdf